CLINICAL TRIAL: NCT00315692
Title: Evaluation of a Multiple Biomarker Assay to Estimate the Risk of Ovarian Cancer in Patients Presenting With a Pelvic Mass.
Brief Title: Risk of Ovarian Cancer in Patients With a Pelvic Mass
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-03 Pelvic Mass Study
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Premenopausal women
  Interventions: Device: Biomarker Assay (CA125 and HE4)
- Postmenopausal women
  Interventions: Device: Biomarker Assay (CA125 and HE4)

INTERVENTIONS:
Device: Biomarker Assay (CA125 and HE4)

SUMMARY:
The purpose of this clinical trial is to evaluate the ability of multiple serum biomarkers to estimate the risk of ovarian cancer in women presenting with pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass).

DETAILED DESCRIPTION:
The Pelvic Mass study is a prospective, multi-center, double blind, statistically powered clinical trial that will enroll female subjects ≥18 years of age presenting to a gynecologist or gynecological oncologist with a pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass) who are scheduled to undergo surgery.

The serum tumor marker CA125 has been the most widely used marker in ovarian cancer, however, it is not sufficiently sensitive or specific for the detection of early stage disease. The levels of soluble mesothelin related peptides (SMRP) and HE4 have also recently been found to be elevated in women with ovarian cancer. The results of a pilot study suggest that the use of HE4 may improve the sensitivity of CA125 and provide for stratification of patients presenting with a pelvic mass into high, intermediate and low risk groups.

HE4 and CA125 serum levels will be evaluated in this study for their ability to stratify patients presenting with a pelvic mass into risk groups with low, intermediate or high probabilities of harboring an ovarian cancer at the time of initial presentation. The algorithm using these two serum markers to stratify patients that was developed using pilot study data will be evaluated in this prospective multicenter pelvic mass study. We will also evaluate the inclusion of additional biomarkers and risk factors, such as ultrasound score, age, and menopausal status, into the algorithm to see if there is any improvement in the stratification of patients into the risk groups.

The primary objective of the study is to estimate the risk of finding ovarian cancer at the time of surgery in pre- and post-menopausal women presenting with pelvic mass. Multiple serum biomarkers (CA125 and HE4) will be evaluated to estimate the risk that the patient is harboring an ovarian cancer at the time of presentation.

The secondary objective of the study is to develop a multivariate predictive algorithm combining CA125 and HE4 with radiological imaging results, and patient risk factors (such as age, menopausal status and ethnicity) to estimate the risk of ovarian cancer, including low malignant potential (LMP) / borderline tumors, at the time of surgery in patients presenting with a pelvic mass.

The exploratory endpoints will include the evaluation of serum, plasma and/or urine levels of CA125, HE4 and other additional novel biomarkers such as SMRP, alone and in combination with radiological imaging results and subject risk factors to determine their ability to estimate the risk of cancer at the time of surgery in patients presenting with a pelvic mass.

ELIGIBILITY:
Inclusion Criteria:

* Females selected to undergo laparotomy or laparoscopy based on a finding of pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass);
* Pre- and post-menopausal women greater than or equal to 18 years of age;
* Pelvic mass must be demonstrated by ultrasound
* Able to understand and sign Informed Consent

Exclusion Criteria:

* Treatment for any malignancy (with the exception of non-melanoma skin cancer) within the last five years
* Subjects receiving cytotoxic chemotherapies, such as cyclophosphamide or methotrexate
* Subjects with previous bilateral oophorectomy
* Any subject known to be pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing surgery for the removal of a pelvic mass.
Sampling Method: Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2005-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Cancer vs Benign Disease

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moore, M.D., Principal Investigator — Womens and Infant's Hosapital of Rhode Island
Locations (2):
- United States (2):
  - Fujirebio Diagnostics, Inc, Malvern, Pennsylvania
  - Richard Moore, Providence, Rhode Island

REFERENCES:
- [Derived] Moore RG, McMeekin DS, Brown AK, DiSilvestro P, Miller MC, Allard WJ, Gajewski W, Kurman R, Bast RC Jr, Skates SJ. A novel multiple marker bioassay utilizing HE4 and CA125 for the prediction of ovarian cancer in patients with a pelvic mass. Gynecol Oncol. 2009 Jan;112(1):40-6. doi: 10.1016/j.ygyno.2008.08.031. Epub 2008 Oct 12. PMID 18851871